CLINICAL TRIAL: NCT07349342
Title: Comparative Effects of Stable Versus Unstable Resistance Training on Lipid Profile Selected Physical Fitness and Renal Biomarkers of Untrained Male University Students
Brief Title: Stable Versus Unstable Resistance Training Effects on Physical Fitness and Physiological Biomarkers of Untrained Male University Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Cherinet Zewdie Zemela, Principal Investigator, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNS-IRB/05/2015/2023
Record Dates: First submitted 2025-12-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: No Condition; Health Young Males
Keywords: eGFR; urinary albumin to creatinine ratio; lipid profile; muscular strength; body composition; muscle; TRX
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This study employs a randomized pre-post-test experimental design with three groups. It involves a stable and unstable resistance training intervention for two training groups and a control group without training intervention but, advised to continue their regular daily routine.
Masking Description: Participants were randomly assigned to a stable, unstable, and control group by computer software. All participants and the researcher know the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unstable resistance training group (Experimental): Receiving total body resistance exercise (TRX) training intervention
  Interventions: Other: resistance training
- Control group (No Intervention): no any structured exercise training intervention
- stable resistance training group (Experimental): receiving traditional resistance training intervention
  Interventions: Other: resistance training

INTERVENTIONS:
Other: resistance training — stable resistance training is represented by traditional resistance training using equipment like medicine ball, resistance machine and own body mass
  Arms: stable resistance training group
Other: resistance training — TRX based resistance training for the upper, lower and abdominal region muscles
  Arms: Unstable resistance training group

SUMMARY:
The goal of this clinical trial is to learn the effects of stable and unstable resistance training on physical fitness, kidney function and blood lipid tests in healthy young male volunteers. The main questions it aims to answer are:

* Do both stable and unstable resistance training increase the level of urinary protein clearance greater than the control group?
* What is the difference in improvement of lipid profiles among the groups?
* Does unstable resistance training mode rise muscular endurance greater than stable resistance training?

Researchers will compare stable and unstable resistance training to see if there are differences on physical fitness measures, blood lipid and urinary protein tests.

Participants, in their respective group will receive ten weeks of:

* Stable resistance training
* Unstable resistance training or
* No exercise training intervention

DETAILED DESCRIPTION:
This study included volunteer male untrained students living at Kotebe University of Education. Priori statistical power analysis (G*Power version 3.1.9.2, Stuttgart, Germany) was used to estimate the sample size. Based on earlier research, a moderate to high effect size (0.295) was assumed, and considering a dropout probability of 10%, a sample of 54 participants was enough to meet adequate statistical power. All participants provided written informed consent to participate in this study. The training protocol will include ten resistance exercises for each intervention, performed three times a week for 10 weeks. Each session lasts 60 minutes, including a 10 to 15-minute warm-up, a 40-minute main exercise targeting core, upper, and lower limb muscles, and a 5 to 10-minute cool-down and stretching. The protocol will adhere to basic training principles like overload, progression, and specificity. The training will take place in the university gymnasium. The study will be conducted in accordance with local legislation and institutional requirements. It will be strictly governed by the ethical principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* No resistance training within the previous six months
* Completing a written informed consent document
* Responding to the physical activity readiness questionnaire (PAR-Q) and becoming convenient

Exclusion Criteria:

* A history of musculoskeletal injury
* Chronic diseases, including known kidney disease
* A habit of alcohol or drug abuse

Ages: 20 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Urinary Albumin | At baseline and after 10 weeks of resistance training interventions
  * It will be measured using random urine samples in milligrams per liter
  * The minimum value is 0, the maximum is 20
  * A higher score means a worse outcome
Urinary Creatinine | At baseline and after 10 weeks of training intervention
  * It will be measured using random urine samples in millimoles per liter
  * The minimum value is 3, the maximum is 25.
  * A higher score means a better outcome
Urinary albumin to creatinine ratio | At baseline and after 10 weeks of resistance training interventions
  * Urinary albumin to creatinine ratio is computed by dividing the obtained urinary albumin by urinary creatinine
  * It is measured in milligrams per millimole
  * The minimum value is 0, the maximum is 3
  * A high score means a worse outcome
Serum Creatinine | At baseline and after 10 weeks of resistance training intervention
  * It is measured using a fasting blood sample in micromoles per liter
  * The minimum value is 50, the maximum is 110
  * A higher score means a worse outcome
Estimated Glomerular Filtration Rate | At baseline and after 10 weeks of resistance training interventions
  * Estimated glomerular filtration rate is computed using a serum creatinine-based equation
  * The scores are reported in milliliters per minute per 1.73 square meters
  * The minimum value is 90, the maximum is 130
  * A higher score means a better renal function
High-Density Lipoprotein Cholesterol | At baseline and after 10 weeks of resistance training
  * It is measured using a fasting blood sample tests in millimoles per liter
  * The minimum value is 1, the maximum is greater than or equal to 2
  * A higher score means a protective and better outcome
Low-Density Llipoprotein Cholesterol | At baseline and after 10 weeks of resistance training
  * It is measured using a fasting blood sample in millimoles per liter
  * The minimum value is 0, the maximum is 2.6
  * A higher score means a worse outcome
Total Cholesterol | At baseline and after 10 weeks of resistance training
  * It is measured using a fasting blood sample test in millimoles per liter
  * The minimum score is 0, the maximum is 5.2
  * A higher score means a worse outcome
Triglycerides | At baseline and after 10 weeks of resistance training
  * Triglycerides are measured using a fasting blood sample test in millimoles per liter
  * The minimum value is 0, the maximum is 1.7
  * A higher score means a worse outcome
Hand Grip Strength | At baseline and after 10 weeks of training intervention
  * Hand grip strength test will be used to measure muscular strength
  * It is measured in kilograms
  * The minimum value is 27, the maximum is 56
  * A higher score means a better outcome
Muscular Endurance | At baseline and after 10 weeks of training intervention
  * Push-up and sit-up tests will be used to measure muscular endurance
  * The number of repetitions is a unit for both tests
  * The minimum score for push-up is 20, the maximum is 40
  * The minimum value for sit-up is 25, the maximum is 45
  * A higher score means a better outcome
Core Endurance | At baseline and after 10 weeks of training intervention
  * The McGill core endurance test will be conducted and reported in seconds
  * The minimum value is 45, the maximum is 120
  * A higher score means a better outcome
Flexibility | At baseline and after 10 weeks of training intervention
  * Sit and reach test will be conducted and reported in centimeters
  * The minimum value is 20, and the maximum is 35
  * A higher score means a better outcome
Body Fat Percentage | At baseline and after 10 weeks of training intervention
  * It will be estimated using 3 site skin fold measures in millimeters
  * Body density will be calculated by the Jackson & Pollock equation
  * The obtained density is converted into body fat percentage using the Sir equation
  * The minimum value is 10, the maximum is 22
  * A higher score means aworse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aschenaki T Tessema, Ph.D., Study Chair — Addis Ababa University; Cherinet Z Zemela, MSc, Principal Investigator — Kotebe University of Education; Zeru B Tola, Ph.D., Study Chair — Addis Ababa University
Locations (1):
- Kotebe University of Education, Addis Ababa, Yeka Sub City, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
After publication on journals, I will share all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning one year after publication and ending 2 years after the publication
Access Criteria: data will be shared with reasonable request from any researcher who brings proposed analysis.